CLINICAL TRIAL: NCT06762886
Title: Aerobic Exercises Versus Laser Puncture Therapy on Immune Response Following Neck Lymph Node Dissection
Brief Title: Aerobic Exercises Versus Laser Puncture on Immune Response Following Neck Lymph Node Dissection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Gamal Fawzy El-Sayed, Doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004069
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Neck Lymph Node Dissection; Immune Defects
Keywords: Aerobic Exercises; Laser Puncture Therapy
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Cycle ergometer treatment protocol (Group 1):
  The case was lying back in a comfortable position on the stationary bike ergometer when the exercise test was conducted. The exercise test began with a 3-minute warm-up session of unloaded cycling on a cycle ergometer, and then progressed at a rate of 10 W per minute up to the subject's threshold. After cycling for 30 W to warm up, the intensity was raised by 15 W every 60 seconds until fatigue, after which the individuals cycled for 30 W to cool down. This treatment protocol was administered to each patient 3 times/week for a total of 15 minutes of treatment, broken into intervals of two to three minutes each.
  Low-level laser treatment protocol (Group 2):
  The laser probe was administered using the contact approach on the dorsal midline, in the depression below the spinous process of C7 at Governor Vessel, with the patient seated in a chair with back support (GV - 14 Dazhui). The primary power switch was activated. The following set
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cycle ergometer treatment protocol (Group 1): (Experimental): Twenty cases with decreased white blood cell counts after neck lymph nodes and deficient in blood immunological functions made up this group. They underwent aerobic exercise training on a cycle ergometer. The cases received one 15-minute session, three sessions per week, for two months, with follow-up after the course of treatment
  Interventions: Device: Cycle ergometer
- Low-level laser treatment protocol (Group 2): (Experimental): Twenty cases with underdeveloped blood immune systems; decreased white blood cell counts after having their neck lymph nodes removed, a low-level laser puncture was performed on the Governing Vessel 14 acupuncture point. They received a 15-minute session, three sessions per week, for two months, with follow-up after the course of treatment
  Interventions: Device: Low-level laser therapy

INTERVENTIONS:
Device: Cycle ergometer — The case was lying back in a comfortable position on the stationary bike ergometer when the exercise test was conducted. The exercise test began with a 3-minute warm-up session of unloaded cycling on a cycle ergometer, and then progressed at a rate of 10 W per minute up to the subject's threshold. After cycling for 30 W to warm up, the intensity was raised by 15 W every 60 seconds until fatigue, after which the individuals cycled for 30 W to cool down. This treatment protocol was administered to each patient 3 times/week for a total of 15 minutes of treatment, broken into intervals of two to three minutes each.
  Arms: Cycle ergometer treatment protocol (Group 1):
Device: Low-level laser therapy — The laser probe was administered using the contact approach on the dorsal midline, in the depression below the spinous process of C7 at Governor Vessel, with the patient seated in a chair with back support (GV - 14 Dazhui). The primary power switch was activated. The following settings were used for applying laser puncture: 5 mW, the maximum average power. Type of laser: gallium arsenide (Ga-As), 904 nm wavelength, 5 kHz maximum repetition rate - Program: Maintaining programs for people who had their neck lymph nodes removed and have a low leukocyte count, up to 30 J/cm2 of energy, a 2 J/cm2 energy density, and protective glasses were required to prevent irreversible eye injury from either direct or indirect laser exposure. The treatment took place for 15 minutes.
  Arms: Low-level laser treatment protocol (Group 2):

SUMMARY:
Group (1): Twenty cases with decreased white blood cell counts after neck lymph nodes and deficient in blood immunological functions made up this group. They underwent aerobic exercise training on a cycle ergometer. The cases received one 15-minute session, three sessions per week, for two months, with follow-up after the course of treatment.

Group (2): Twenty cases with underdeveloped blood immune systems; decreased white blood cell counts after having their neck lymph nodes removed, a low-level laser puncture was performed on the Governing Vessel 14 acupuncture point. They received a 15-minute session, three sessions per week, for two months, with follow-up after the course of treatment

DETAILED DESCRIPTION:
Inclusion criteria:

All cases were checked carefully by a physician before the study procedures. All cases were approximately the same age. All cases were conscious. All cases in both groups obtained the same medications and they received three sessions per week for 2 months. All patients enrolled in the study had a deficiency in blood immune functions post neck lymph node dissection and received chemotherapy.

Exclusion criteria:

Patients with associated disease (other pathological conditions), patients suffering from metastases, patients taking medications that alter leukocytes count and pregnancy or epilepsy.

Measurement procedures:

The total number of circulating leukocytes (white blood cells) and the differential lymphocyte count were adopted in the current academic work to measure the immunological response in both groups. These were carried out two months after the start of treatment and before the first session: pre-treatment application and post-treatment after two months. The measurement steps were as follows:

Measurement of immune response:

The cases were seated when immune response was measured. Morning peripheral blood sample aspiration was followed by venous blood collection into sterile glass containers with the necessary anticoagulants and preservatives. A Coulter hematology analyzer (Coulter Electronics, USA) was used to perform differential counts of lymphocytes and the total leukocyte count.

Treatment procedures: The following steps were adopted to complete the treatment procedures: When a patient comes in for treatment, they were given a thorough explanation of the procedures' goals as well as their physiological and therapeutic advantages.

Cycle ergometer treatment protocol (Group 1):

The case was lying back in a comfortable position on the stationary bike ergometer when the exercise test was conducted. The exercise test began with a 3-minute warm-up session of unloaded cycling on a cycle ergometer, and then progressed at a rate of 10 W per minute up to the subject's threshold. After cycling for 30 W to warm up, the intensity was raised by 15 W every 60 seconds until fatigue, after which the individuals cycled for 30 W to cool down. This treatment protocol was administered to each patient 3 times/week for a total of 15 minutes of treatment, broken into intervals of two to three minutes each.

Low-level laser treatment protocol (Group 2):

The laser probe was administered using the contact approach on the dorsal midline, in the depression below the spinous process of C7 at Governor Vessel, with the patient seated in a chair with back support (GV - 14 Dazhui). The primary power switch was activated. The following settings were used for applying laser puncture: 5 mW, the maximum average power. Type of laser: gallium arsenide (Ga-As), 904 nm wavelength, 5 kHz maximum repetition rate - Program: Maintaining programs for people who had their neck lymph nodes removed and have a low leukocyte count, up to 30 J/cm2 of energy, a 2 J/cm2 energy density, and protective glasses were required to prevent irreversible eye injury from either direct or indirect laser exposure. The treatment took place for 15 minutes.

ELIGIBILITY:
Inclusion Criteria:

* All cases were checked carefully by a physician before the study procedures. All cases were approximately the same age.

All cases were conscious. All cases in both groups obtained the same medications and they received three sessions per week for 2 months.

All patients enrolled in the study had a deficiency in blood immune functions post neck lymph node dissection and received chemotherapy.

Exclusion Criteria:

* Patients with associated disease (other pathological conditions). patients suffering from metastases. patients taking medications that alter leukocytes count and pregnancy or epilepsy.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Leukocyte total count and differential lymphocyte count measurements | 2 months
  Measurement of immune response:
  The cases were seated when immune response was measured. Morning peripheral blood sample aspiration was followed by venous blood collection into sterile glass containers with the necessary anticoagulants and preservatives. A Coulter hematology analyzer (Coulter Electronics, USA) was used to perform differential counts of lymphocytes and the total leukocyte count.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Giza, Egypt